CLINICAL TRIAL: NCT03073733
Title: A Prospective, Multicenter, Randomized, Study of the Safety and Efficacy of Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects With Retinitis Pigmentosa (RP)
Brief Title: Safety and Efficacy of Intravitreal Injection of Human Retinal Progenitor Cells in Adults With Retinitis Pigmentosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: jCyte, Inc (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JC-02
Record Dates: First submitted 2017-03-02; First posted 2017-03-08 (Actual); Results first posted 2022-01-21 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects, their family members and clinical staff performing key efficacy assessments will be masked to the randomization assignment of subjects. Due to the nature of some safety assessments and the sham treatment, not all personnel can be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Test (jCell injection) dose level 1 (Experimental): single intravitreal injection of 3.0 x 10e6 human retinal progenitor cells into the eye with the poorest visual acuity or, if vision is comparable in both eyes, the non-dominant eye
  Interventions: Biological: human retinal progenitor cells
- Sham treated Control (Other): a mock injection will be performed on the eye with the poorest vision in each Control subject (designated as the "study eye")
  Interventions: Other: Mock injection
- test (jCell injection) dose level 2 (Experimental): single intravitreal injection of 6.0 x 10e6 human retinal progenitor cells into the eye with the poorest visual acuity or, if vision is comparable in both eyes, the non-dominant eye
  Interventions: Biological: human retinal progenitor cells

INTERVENTIONS:
Biological: human retinal progenitor cells — live suspension of 3.0 or 6.0 x 10e6 human retinal progenitor cells (hRPC) suspended in clinical grade medium injected intravitreally under local anesthesia
  Other Names: jCell
  Arms: Test (jCell injection) dose level 1; test (jCell injection) dose level 2
Other: Mock injection — pressing the hub of a syringe with no needle against the eye to mimic intravitreal injection
  Arms: Sham treated Control

SUMMARY:
This study evaluates the changes in visual function at 12 months following a single injection of human retinal progenitor cells compared to sham treated controls in a cohort of adult subjects with RP.

DETAILED DESCRIPTION:
There is no effective treatment for RP; once photoreceptors are lost, they do not regenerate. The rate of deterioration of vision varies from person to person, with most people with RP legally blind by age 40. Preclinical studies demonstrated that transplantation of retinal progenitor cells into the eye can result in both photoreceptor replacement and significant slowing of host photoreceptor loss. Thus, the primary goal of this therapy is to preserve, and potentially improve, vision by intervening in the disease at a time when dystrophic host photoreceptors can be protected and reactivated. Based on the demonstration of acceptable safety and tolerability in a phase 1/2a study, this phase 2b study is designed as a controlled comparison of the changes in visual function and functional vision in subjects who receive a single jCell injection in comparison to a comparable sham-treated control group of subjects with RP.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of RP confirmed by ERG and willing to consent to mutation typing, if not already done Best corrected visual acuity (BCVA) 20/80 or worse and no worse than 20/800 Adequate organ function and negative infectious disease screen Female of childbearing potential must have negative pregnancy test and be willing to use medically accepted methods of contraception throughout the study

Exclusion Criteria:

Eye disease other than RP that impairs visual function Pseudo-RP, cancer-associated retinopathies History of malignancy or other end-stage organ disease, or any chronic disease requiring continuous treatment with system steroids, anticoagulants or immunosuppressive agents Known allergy to penicillin or streptomycin Treatment with corticosteroids or any investigational or neuroprotectant therapy within 90 days of enrollment Cataract surgery within 3 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitul Mehta, MD, Principal Investigator — UCI; David Liao, MD, Principal Investigator — RVA; Anthony Joseph, MD, Principal Investigator — OCB
Locations (3):
- United States (3):
  - Gavin Herbert Eye Inst, Univ Cal Irvine, Irvine, California
  - Retina-Vitreous Associates Medical Group, Los Angeles, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 85 subjects were enrolled; 84 subjects were randomized
Pre-assignment Details: One subject received a 4.0 x 10e6 dose prior to a major protocol amendment that excluded this dose group; this subject is not included in the analyses presented.
Groups:
- Sham Treated Control: Mock injection: pressing the hub of a syringe with no needle against the study eye to mimic intravitreal injection.
- Test (jCell Injection) Dose Level 1: Single intravitreal injection of 3.0 x 10e6 retinal progenitor cells into the study eye
- Test (jCell Injection) Dose Level 2: Single intravitreal injection of 6.0 x 10e6 retinal progenitor cells into the study eye
Period: Overall Study
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Started | 29 | 27 | 27
Completed | 28 | 26 | 26
Not Completed | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject received 4M dose prior to major protocol amendment that excluded this dose group; this subject is not included in the presented analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2 | Total
Number analyzed (Participants) | 29 | 27 | 27 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 24 | 71
  >=65 years | 6 | 3 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 15 | 13 | 35
  Male | 22 | 12 | 14 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 7 | 16
  Not Hispanic or Latino | 24 | 23 | 20 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 2 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 22 | 23 | 20 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 27 | 83
Selection of study eye [Count of Participants; unit: Participants]
  study eye OD | 12 | 12 | 14 | 38
  study eye OS | 17 | 15 | 13 | 45

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity (BCVA)
Description: Mean change in BCVA in study eye from baseline to month 12 as assessed by E-ETDRS in ITT population. A letter score is used to compare change over time, with a higher number of letters representing better visual function, and a lower number of letters representing worse visual function. For example, 85 letters is equivalent to 20/20 visual acuity and 5 letters is equivalent to 20/800 visual acuity. A change value is derived for each subject by taking the letter score at 12 months and subtracting the letter score at baseline. A mean of all change values is then calculated for each arm.
Time Frame: 12 months
Population: ITT: All randomized subjects who provide any post-randomization data. One subject received a 4.0 x 10e6 dose prior to a protocol amendment that excluded this dose level; this subject is not included in these analyses. Also, of the 83 remaining subjects to be enrolled and randomized, 80 completed the study.
Measure: Mean (Standard Deviation); unit: Letters correct
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 28 | 26 | 26
Letters correct | 3.9 (9.92) | 1.3 (14.14) | 2.6 (21.53)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 1; Test type: Superiority; p = 0.582, linear model for repeated measures; least squares mean difference = -2.2, 95% CI 2-sided [-10.3 to 5.8], Standard Error of Mean 2.90
Statistical Analysis 2: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.984, linear model for repeated measures; least squares mean difference = -0.1, 95% CI 2-sided [-8.2 to 8.0], Standard Error of Mean 2.91

2. Secondary Outcome: Contrast Sensitivity (CS) at 1.0 CPD
Description: Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. For example, if a subject's CS peak appears to be at 2.0 CPD, then additional testing occurs at 1.0 and 4.0 CPD. RP patients have suppressed CS curves and the most common pattern widths are at 0.5, 1.0, 2.0, and 4.0 CPD. Severely impaired subjects (e.g., BCVA < 20/400) usually have flat curves with low values (e.g., 1.28), while in mildly impaired RP subjects the values can be higher (e.g., 7.12), but are rarely near normal. These data represent mean change in CS from baseline to 12 months, with greater values representing greater improvement in visual function.
Time Frame: 12 months
Population: mITT: all randomized subjects who provide any post-randomization data, excluding subjects with missing baseline or who are below the limit of detection (LOD) at baseline; shown here are subjects who could be assessed at a pattern width of 1.0 CPD, which applies to the largest number of participating subjects as compared to the other CPD pattern widths.
Measure: Mean (Standard Deviation); unit: CS at 1.0 cycles per degree (CPD)
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 21 | 19 | 24
CS at 1.0 cycles per degree (CPD) | 0.4331 (1.5011) | 1.9145 (4.3072) | 0.1142 (4.9526)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 1; Test type: Superiority; p = 0.290, linear model for repeated measures; least squares mean difference = 1.2986, 95% CI 2-sided [-1.1341 to 3.7313], Standard Error of Mean 0.8744
Statistical Analysis 2: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.759, linear model for repeated measures; least squares mean difference = -0.3542, 95% CI 2-sided [-2.6516 to 1.9433], Standard Error of Mean 0.7793

3. Secondary Outcome: Kinetic Visual Field (KVF)
Description: Mean change in total area (degrees squared) of all islands of vision from baseline to 12 months.
Time Frame: 12 months
Population: mITT: all randomized subjects who provide any post-randomization data, excluding subjects with missing baseline or who are below the limit of detection (LOD) at baseline.
Measure: Mean (Standard Deviation); unit: Total area (degrees squared)
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 28 | 26 | 25
Total area (degrees squared) | 260.19 (900.024) | -44.02 (1001.614) | 560.19 (2453.259)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 1; Test type: Superiority; p = 0.515, linear model for repeated measures; least squares mean difference = -278.73, 95% CI 2-sided [-1126.21 to 568.75], Standard Error of Mean 305.192
Statistical Analysis 2: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.499, linear model for repeated measures; least squares mean difference = 292.18, 95% CI 2-sided [-562.87 to 1147.23], Standard Error of Mean 308.659

4. Secondary Outcome: Low Luminance Mobility Test (LLMT)
Description: The LLMT identifies the performance of RP patients as they walk along an indoor pathway of arrows and obstacles at varying lighting levels. The Critical Illumination Level (CIL) is the light level below which the patient has a markedly slower pace and more errors than all light levels above (brighter than) that point. The LLMT uses light levels that go from very dim (0.12 lux) to a bright indoor room (500 lux), with evenly spaced increments that increase light by doubling the brightness of the room from the prior level. These evenly spaced light levels have been converted to a scale score to enable easier calculation of change scores. The dimmest light level of 0 lux (completely dark room) corresponds to a scale score of 13, whereas the brightest light level of 500 lux corresponds to a scale score of 0. A positive scale score change from baseline to 12 months represents improvement in low light vision, whereas a negative scale score change represents a decline in low light vision.
Time Frame: 12 months
Population: Modified ITT: all randomized subjects who provide any post-randomization data, excluding subjects with missing baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 24 | 25 | 24
Scores on a scale | 0.6 (2.00) | -0.3 (2.49) | 0.2 (1.96)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 1; Test type: Superiority; p = 0.160, linear model for repeated measures; least squares mean difference = -0.9, 95% CI 2-sided [-2.1 to 0.3], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.622, linear model for repeated measures; least squares mean difference = -0.3, 95% CI 2-sided [-1.5 to 0.9], Standard Error of Mean 0.43

5. Secondary Outcome: Low Vision Functional Questionnaire (Visual Ability)
Description: The VA LV VFQ-48 (VFQ) is used to capture changes in patients' self-reporting of their difficulty with reading, mobility and performing other daily living activities affected by visual impairment. There are 4 scales on the VFQ including Visual Information, Reading, Visual Motor, and Mobility. A fifth value, Visual Ability, is an aggregate score of the 4 scales, measured in units called logits, and is calculated for each person based on item weighting using Raasch analysis. Visual Ability is used broadly to represent changes in subject-reported outcomes from visit to visit. Higher positive values on the Visual Ability score represent better function and less impairment, whereas lower or negatives scores represent worse function or more impairment. Change in the Visual Ability scale on the VFQ is calculated by taking a subject's score at 12 months and subtracting from it the baseline score.
Time Frame: 12 months
Population: mITT: all randomized subjects who provide any post-randomization data, excluding subjects with missing baseline.
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 28 | 26 | 26
logits | 0.225 (0.4194) | 0.146 (0.5228) | 0.360 (0.6963)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 1; Test type: Superiority; p = 0.442, linear model for repeated measures; least squares mean difference = -0.111, 95% CI 2-sided [-0.399 to 0.176], Standard Error of Mean 0.1038
Statistical Analysis 2: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.401, linear model for repeated measures; least squares mean difference = 0.122, 95% CI 2-sided [-0.165 to 0.409], Standard Error of Mean 0.1037

6. Secondary Outcome: Safety of Intravitreal Injection of Retinal Progenitor Cells (RPC)
Description: Assessed by treatment emergent adverse events, immunogenicity and safety visual assessments
Time Frame: 12 months
Population: Safety population: all subjects who receive any study treatment (including sham); subjects who did not complete may not have data at 12-month time point
Measure: Number; unit: participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 29 | 27 | 27
participants
  Subjects with TEAE | 15 | 20 | 21
  Subjects with related/possibly related TEAE | 7 | 14 | 13
  Subjects with severe TEAE | 0 | 3 | 1
  Subjects with SAE | 0 | 1 | 0
  Subjects with CME absent at baseline and present at M12 (OCT) | 1 | 0 | 0
  Subjects with clinically significant abnormal conjunctiva absent at baseline and present at M12 | 0 | 2 | 0
  Subjects with clinically significant abnormal sclera absent at baseline and present at M12 | 0 | 1 | 0
  Subjects with clinically significant abnormal AC flare absent at baseline and present at M12 | 0 | 0 | 0

7. Post Hoc Outcome: Responder Analysis (≥10 Letters): Best Corrected Visual Acuity (BCVA) - PP Population
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population (N=76), with a responder being defined as someone who gains at least 10 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. The PP population excludes seven subjects with major protocol violations, including two subjects who received a different treatment than the group to which they were randomized, four subjects with preexisting ophthalmic conditions meeting exclusion criteria (three glaucoma and one amblyopia), and one subject who experienced an intraocular lens subluxation (i.e., the displacement of a replacement lens following previous cataract surgery - unrelated to study drug) and could not perform endpoint testing at 12 months.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 26 | 25 | 23
Participants | 5 | 4 | 9
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.205, Fisher Exact

8. Post Hoc Outcome: Responder Analysis (≥13 Letters): Best Corrected Visual Acuity (BCVA) - PP Population
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population (N=76), with a responder being defined as someone who gains at least 13 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. The PP population excludes seven subjects with major protocol violations, including two subjects who received a different treatment than the group to which they were randomized, four subjects with preexisting ophthalmic conditions meeting exclusion criteria (three glaucoma and one amblyopia), and one subject who experienced an intraocular lens subluxation (i.e., the displacement of a replacement lens following previous cataract surgery - unrelated to study drug) and could not perform endpoint testing at 12 months.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 26 | 25 | 23
Participants | 3 | 4 | 7
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.157, Fisher Exact

9. Post Hoc Outcome: Responder Analysis (≥15 Letters): Best Corrected Visual Acuity (BCVA) - PP Population
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population (N=76), with a responder being defined as someone who gains at least 15 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. The PP population excludes seven subjects with major protocol violations, including two subjects who received a different treatment than the group to which they were randomized, four subjects with preexisting ophthalmic conditions meeting exclusion criteria (three glaucoma and one amblyopia), and one subject who experienced an intraocular lens subluxation (i.e., the displacement of a replacement lens following previous cataract surgery - unrelated to study drug) and could not perform endpoint testing at 12 months.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 26 | 25 | 23
Participants | 2 | 3 | 6
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.125, Fisher Exact

10. Post Hoc Outcome: Responder Analysis (≥20 Letters): Best Corrected Visual Acuity (BCVA) - PP Population
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population (N=76), with a responder being defined as someone who gains at least 20 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. The PP population excludes seven subjects with major protocol violations, including two subjects who received a different treatment than the group to which they were randomized, four subjects with preexisting ophthalmic conditions meeting exclusion criteria (three glaucoma and one amblyopia), and one subject who experienced an intraocular lens subluxation (i.e., the displacement of a replacement lens following previous cataract surgery - unrelated to study drug) and could not perform endpoint testing at 12 months.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 26 | 25 | 23
Participants | 1 | 2 | 4
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.173, Fisher Exact

11. Post Hoc Outcome: Best Corrected Visual Acuity (BCVA) - PP Population
Description: Mean change in BCVA in study eye from baseline to month 12 as assessed by E-ETDRS in the Per Protocol (PP) population (N=76). The PP population excludes seven subjects with major protocol violations, including two subjects who received a different treatment than the group to which they were randomized, four subjects with preexisting ophthalmic conditions meeting exclusion criteria (three glaucoma and one amblyopia), and one subject who experienced an intraocular lens subluxation (i.e., the displacement of a replacement lens following previous cataract surgery - unrelated to study drug) and could not perform endpoint testing at 12 months. Refer to Outcome Measure #1 for more information on how change in BCVA from baseline to month 12 is assessed.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study
Measure: Mean (Standard Deviation); unit: Letters correct
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 26 | 25 | 23
Letters correct | 2.8 (8.69) | 3.0 (11.43) | 7.4 (15.57)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.099, t-test, 1 sided; Pooled t-test (variance ratio of 3.2)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.130, t-test, 1 sided; Pooled t-test (variance ratio of 1.9)

12. Post Hoc Outcome: Responder Analysis (≥100%): Peak Contrast Sensitivity (CS) - PP Population
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population (N=76), with a responder being defined as someone who gains at least 100% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to month 12 is assessed.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study, of which 65 posted a measurable CS value at both baseline and 12 months. Missing values were not imputed for purposes of the PP Population analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 23 | 20 | 22
Participants | 1 | 2 | 5
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.0959, Fisher Exact

13. Post Hoc Outcome: Responder Analysis (≥150%): Peak Contrast Sensitivity (CS) - PP Population
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population (N=76), with a responder being defined as someone who gains at least 150% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to month 12 is assessed.
Time Frame: 12 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 23 | 20 | 22
Participants | 1 | 0 | 4
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.1868, Fisher Exact

14. Post Hoc Outcome: Responder Analysis (≥200%): Peak Contrast Sensitivity (CS) - PP Population
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population (N=76), with a responder being defined as someone who gains at least 200% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to month 12 is assessed.
Time Frame: 12 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 23 | 20 | 22
Participants | 1 | 0 | 2
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.608, Fisher Exact

15. Post Hoc Outcome: Peak Contrast Sensitivity (CS) - PP Population
Description: Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. The data shown here are for mean change from baseline to 12 months in the peak of the CS curve in the Per Protocol (PP) population (N=76). Refer to Outcome Measure #7 for background information on the PP population. Refer to Outcome Measure #2 for more information on how change in CS from baseline to month 12 is assessed.
Time Frame: 12 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Peak CS
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 23 | 20 | 22
Peak CS | 1.3454 (4.4164) | 0.1294 (2.4379) | 3.1329 (12.4076)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.264, t-test, 1 sided; Unpooled t-test (variance ratio of 7.9)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.139, t-test, 1 sided; Unpooled t-test (variance ratio of 25.9)

16. Post Hoc Outcome: Kinetic Visual Field (KVF) - PP Population
Description: Mean change in total area (degrees squared) of all islands of vision from baseline to 12 months in the Per Protocol (PP) Population (N=76). Refer to Outcome Measure #7 for background information on the PP population.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study.
Measure: Mean (Standard Deviation); unit: Total area (degrees squared)
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 26 | 25 | 23
Total area (degrees squared) | 229.13 (908.525) | -37.81 (1021.757) | 594.47 (2558.858)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.261, t-test, 1 sided; Unpooled t-test (variance ratio of 7.9)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.139, t-test, 1 sided; Unpooled t-test (variance ratio of 6.3)

17. Post Hoc Outcome: Low Luminance Mobility Test (LLMT) - PP Population
Description: The LLMT identifies the performance of RP patients as they walk along an indoor pathway of arrows and obstacles at varying lighting levels. The Critical Illumination Level (CIL) is the light level below which the patient has a markedly slower pace and more errors than all light levels above (brighter than) that point. The LLMT uses light levels that go from very dim (0.12 lux) to a very bright (500 lux), with evenly spaced increments that increase light by doubling the brightness of the room from the prior level. These evenly spaced light levels have been converted to a scale score to enable easier calculation of change scores. The dimmest level of 0 lux corresponds to a scale score of 13, whereas the brightest level of 500 lux corresponds to a scale score of 0. A positive scale score change from baseline to 12 months represents improvement, whereas a negative scale score change represents a decline. Refer to Outcome Measure #7 for background information on the PP population.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study, of which 66 posted a measurable CIL value at both baseline and 12 months. Missing values were not imputed for purposes of the PP Population analyses.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 22 | 22 | 22
Scores on a scale | 0.6 (2.06) | 0.4 (1.14) | 0.4 (1.82)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.350, t-test, 1 sided; Pooled t-test (variance ratio of 0.8)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.500, t-test, 1 sided; Pooled t-test (variance ratio of 2.5)

18. Post Hoc Outcome: Low Vision Functional Questionnaire (Visual Ability) - PP Population
Description: The VA LV VFQ-48 (VFQ) is used to capture changes in patients' self-reporting of their difficulty with reading, mobility and performing other daily living activities affected by visual impairment. There are 4 scales on the VFQ including Visual Information, Reading, Visual Motor, and Mobility. A fifth value, Visual Ability, is an aggregate score of the 4 scales, measured in units called logits, and is calculated for each person based on item weighting using Raasch analysis. Visual Ability is used broadly to represent changes in subject-reported outcomes from visit to visit. Higher positive values on the Visual Ability score represent better function and less impairment, whereas lower or negatives scores represent worse function or more impairment. Change in the Visual Ability scale on the VFQ is calculated by taking a subject's score at 12 months and subtracting from it the baseline score. Refer to Outcome Measure #7 for background information on the PP population.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 26 | 25 | 23
logits | 0.238 (0.4324) | 0.151 (0.5329) | 0.371 (0.7335)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.220, t-test, 1 sided; Pooled t-test (variance ratio of 2.9)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.119, t-test, 1 sided; Pooled t-test (variance ratio of 1.9)

19. Post Hoc Outcome: Low Vision Functional Questionnaire (Mobility) - PP Population
Description: The VA LV VFQ-48 (VFQ) is used to capture changes in patients' self-reporting of their difficulty with reading, mobility and performing other daily living activities affected by visual impairment. There are 4 scales on the VFQ including Visual Information, Reading, Visual Motor, and Mobility. The data shown in this outcome measure is focused on the fourth scale, Mobility, and is measured in units called logits. Higher positive values on the Mobility score represent better function and less impairment, whereas lower or negatives scores represent worse function or more impairment. Change in the Mobility scale on the VFQ is calculated by taking a subject's score at 12 months and subtracting from it the baseline score.
Time Frame: 12 months
Population: Per Protocol (PP) population - 74 subjects from this population completed the study
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 26 | 25 | 23
logits | 0.024 (0.499) | 0.256 (0.716) | 0.521 (0.813)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.006, t-test, 1 sided; Pooled t-test (variance ratio of 2.7)

20. Post Hoc Outcome: Responder Analysis (≥10 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55), with a responder being defined as someone who gains at least 10 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. The work undertaken to understand what contributed to variability in measurements in the Phase 2b study, combined with the available published literature, has led to the identification of the characteristics of individuals who provide inconsistent/unreliable data. One such characteristic is found in subjects in whom there is a substantial BCVA disparity of more than 15 letters between their study (worse) eye and fellow (better) eye. This disparity has the potential to lead to variable testing results due to the brain's un-suppression of the image from their worse-seeing eye under clinical study monocular test conditions where their dominant eye is covered.
Time Frame: 12 months
Population: Per Protocol (PP) Population with ≤15 letter baseline BCVA disparity between eyes - 54 subjects from this population completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 21 | 17 | 16
Participants | 2 | 2 | 8
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.009, Fisher Exact

21. Post Hoc Outcome: Responder Analysis (≥13 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55), with a responder being defined as someone who gains at least 13 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. The work undertaken to understand what contributed to variability in measurements in the Phase 2b study, combined with the available published literature, has led to the identification of the characteristics of individuals who provide inconsistent/unreliable data. One such characteristic is found in subjects in whom there is a substantial BCVA disparity of more than 15 letters between their study (worse) eye and fellow (better) eye. This disparity has the potential to lead to variable testing results due to the brain's un-suppression of the image from their worse-seeing eye under clinical study monocular test conditions where their dominant eye is covered.
Time Frame: 12 months
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 21 | 17 | 16
Participants | 1 | 2 | 6
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.029, Fisher Exact

22. Post Hoc Outcome: Responder Analysis (≥15 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55), with a responder being defined as someone who gains at least 15 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. The work undertaken to understand what contributed to variability in measurements in the Phase 2b study, combined with the available published literature, has led to the identification of the characteristics of individuals who provide inconsistent/unreliable data. One such characteristic is found in subjects in whom there is a substantial BCVA disparity of more than 15 letters between their study (worse) eye and fellow (better) eye. This disparity has the potential to lead to variable testing results due to the brain's un-suppression of the image from their worse-seeing eye under clinical study monocular test conditions where their dominant eye is covered.
Time Frame: 12 months
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 21 | 17 | 16
Participants | 0 | 1 | 5
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.010, Fisher Exact

23. Post Hoc Outcome: Responder Analysis (≥20 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55), with a responder being defined as someone who gains at least 20 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. The work undertaken to understand what contributed to variability in measurements in the Phase 2b study, combined with the available published literature, has led to the identification of the characteristics of individuals who provide inconsistent/unreliable data. One such characteristic is found in subjects in whom there is a substantial BCVA disparity of more than 15 letters between their study (worse) eye and fellow (better) eye. This disparity has the potential to lead to variable testing results due to the brain's un-suppression of the image from their worse-seeing eye under clinical study monocular test conditions where their dominant eye is covered.
Time Frame: 12 months
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 21 | 17 | 16
Participants | 0 | 0 | 3
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.072, Fisher Exact

24. Post Hoc Outcome: Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Mean change in BCVA from Baseline to month 12 as assessed by E-ETDRS in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55). The work undertaken to understand what contributed to variability in measurements in the Phase 2b study, combined with the available published literature, has led to the identification of the characteristics of individuals who provide inconsistent/unreliable data. One such characteristic is found in subjects in whom there is a substantial BCVA disparity of more than 15 letters between their study (worse) eye and fellow (better) eye. This disparity has the potential to lead to variable testing results due to the brain's un-suppression of the image from their worse-seeing eye under clinical study monocular test conditions where their dominant eye is covered. Refer to Outcome Measure #1 for more information on how change in BCVA from baseline to month 12 is assessed.
Time Frame: 12 months
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Letters correct
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 21 | 17 | 16
Letters correct | 0.86 (6.54) | 0.82 (7.98) | 10.25 (15.91)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.019, t-test, 1 sided; Unpooled t-test (variance ratio of 5.9)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.019, t-test, 1 sided; Pooled t-test (variance ratio of 3.98)

25. Post Hoc Outcome: Responder Analysis (≥100%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55), with a responder being defined as someone who gains at least 100% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: Per Protocol (PP) Population with ≤15 letter baseline BCVA disparity between eyes - 54 subjects from this population completed the study, of which 45 posted a measurable CS value at both baseline and 12 months. Missing values were not imputed for purposes of this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 18 | 12 | 15
Participants | 0 | 2 | 5
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.013, Fisher Exact

26. Post Hoc Outcome: Responder Analysis (≥150%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55), with a responder being defined as someone who gains at least 150% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 18 | 12 | 15
Participants | 0 | 0 | 4
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.033, Fisher Exact

27. Post Hoc Outcome: Responder Analysis (≥200%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55), with a responder being defined as someone who gains at least 200% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 18 | 12 | 15
Participants | 0 | 0 | 2
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.199, Fisher Exact

28. Post Hoc Outcome: Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. The data shown here are for mean change from baseline to 12 months in the peak of the CS curve in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55). Refer to Outcome Measure #12 for background information on this analysis population. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Peak CS
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 18 | 12 | 15
Peak CS | 0.61 (1.85) | 0.11 (2.76) | 6.09 (13.87)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.075, t-test, 1 sided; Unpooled t-test (variance ratio of 56.3)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.062, t-test, 1 sided; Unpooled t-test (variance ratio of 25.2)

29. Post Hoc Outcome: Kinetic Visual Field (KVF) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: Mean change in total area (degrees squared) of all islands of vision from baseline to 12 months in the Per Protocol (PP) Population with a study eye that is ≤15 letters worse than the fellow eye at baseline (N=55). Refer to Outcome Measure #12 for background information on this analysis population.
Time Frame: 12 months
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Total area (degrees squared)
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 21 | 17 | 16
Total area (degrees squared) | 313.33 (964.08) | -173.46 (1027.19) | 843.93 (3035.82)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.255, t-test, 1 sided; Unpooled t-test (variance ratio of 9.9)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.109, t-test, 1 sided; Unpooled t-test (variance ratio of 8.7)

30. Post Hoc Outcome: Low Luminance Mobility Test (LLMT) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes
Description: The LLMT identifies the performance of RP patients as they walk along an indoor pathway of arrows and obstacles at varying lighting levels. The Critical Illumination Level (CIL) is the light level below which the patient has a markedly slower pace and more errors than all light levels above (brighter than) that point. The LLMT uses light levels that go from very dim (0.12 lux) to very bright (500 lux), with evenly spaced increments that increase light by doubling the brightness of the room from the prior level. These evenly spaced light levels have been converted to a scale score to enable easier calculation of change scores. The dimmest level of 0 lux corresponds to a scale score of 13, whereas the brightest level of 500 lux corresponds to a scale score of 0. A positive scale score change from baseline to 12 months represents improvement, whereas a negative scale score change represents a decline. Refer to Outcome Measure #12 for background information on this analysis population.
Time Frame: 12 months
Population: Per Protocol (PP) Population with ≤15 letter baseline BCVA disparity between eyes - 54 subjects from this population completed the study, of which 46 posted a measurable CIL value at both baseline and 12 months. Missing values were not imputed for purposes of this analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 17 | 14 | 15
scores on a scale | 0.82 (2.24) | 0.43 (1.22) | 0.80 (1.93)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.488, t-test, 1 sided; Pooled t-test (variance ratio of 0.7)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.273, t-test, 1 sided; Pooled t-test (variance ratio of 2.5)

31. Post Hoc Outcome: Responder Analysis (≥10 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye and with the ability to maintain fixation at baseline (N=42), with a responder being defined as someone who gains at least 10 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. Beyond the BCVA disparity characteristic described in the previous post-hoc outcome measures, another characteristic that was found to lead to high degrees of testing variability was the inability to maintain fixation as assessed by a fixation score of 1 on kinetic visual field testing. This inability was due to either an atypical form of RP which caused the development of a central scotoma (blind spot), or the absence of remaining central visual field. These individuals tended to have extremely variable results that were dependent upon their ability to use unsteady "peripheral" eccentric viewing to perform the clinical endpoint tests.
Time Frame: 12 months
Population: Per Protocol (PP) Population with ≤15 letter baseline BCVA disparity between eyes and ability to maintain fixation - 41 subjects from this population completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 14 | 14 | 13
Participants | 1 | 1 | 8
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.004, Fisher Exact

32. Post Hoc Outcome: Responder Analysis (≥13 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye and with the ability to maintain fixation at baseline (N=42), with a responder being defined as someone who gains at least 13 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. Beyond the BCVA disparity characteristic described in the previous post-hoc outcome measures, another characteristic that was found to lead to high degrees of testing variability was the inability to maintain fixation as assessed by a fixation score of 1 on kinetic visual field testing. This inability was due to either an atypical form of RP which caused the development of a central scotoma (blind spot), or the absence of remaining central visual field. These individuals tended to have extremely variable results that were dependent upon their ability to use unsteady "peripheral" eccentric viewing to perform the clinical endpoint tests.
Time Frame: 12 months
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 14 | 14 | 13
Participants | 0 | 1 | 6
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.006, Fisher Exact

33. Post Hoc Outcome: Responder Analysis (≥15 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye and with the ability to maintain fixation at baseline (N=42), with a responder being defined as someone who gains at least 15 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. Beyond the BCVA disparity characteristic described in the previous post-hoc outcome measures, another characteristic that was found to lead to high degrees of testing variability was the inability to maintain fixation as assessed by a fixation score of 1 on kinetic visual field testing. This inability was due to either an atypical form of RP which caused the development of a central scotoma (blind spot), or the absence of remaining central visual field. These individuals tended to have extremely variable results that were dependent upon their ability to use unsteady "peripheral" eccentric viewing to perform the clinical endpoint tests.
Time Frame: 12 months
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 14 | 14 | 13
Participants | 0 | 1 | 5
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.016, Fisher Exact

34. Post Hoc Outcome: Responder Analysis (≥20 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye and with the ability to maintain fixation at baseline (N=42), with a responder being defined as someone who gains at least 20 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. Beyond the BCVA disparity characteristic described in the previous post-hoc outcome measures, another characteristic that was found to lead to high degrees of testing variability was the inability to maintain fixation as assessed by a fixation score of 1 on kinetic visual field testing. This inability was due to either an atypical form of RP which caused the development of a central scotoma (blind spot), or the absence of remaining central visual field. These individuals tended to have extremely variable results that were dependent upon their ability to use unsteady "peripheral" eccentric viewing to perform the clinical endpoint tests.
Time Frame: 12 months
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 14 | 14 | 13
Participants | 0 | 0 | 3
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.098, Fisher Exact

35. Post Hoc Outcome: Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Mean change in BCVA in study eye from baseline to month 12 as assessed by E-ETDRS in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye and with the ability to maintain fixation at baseline (N=42). Beyond the BCVA disparity characteristic described in the previous post-hoc outcome measures, another characteristic that was found to lead to high degrees of testing variability was the inability to maintain fixation as assessed by a fixation score of 1 on kinetic visual field testing. This inability was due to either an atypical form of RP which caused the development of a central scotoma (blind spot), or the absence of remaining central visual field. These individuals tended to have extremely variable results that were dependent upon their ability to use unsteady "peripheral" eccentric viewing to perform the clinical endpoint tests. Refer to Outcome Measure #1 for more information on how change in BCVA from baseline to month 12 is assessed.
Time Frame: 12 months
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Letters correct
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 14 | 14 | 13
Letters correct | 2.00 (5.75) | 0.29 (7.56) | 13.00 (16.47)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.019, t-test, 1 sided; Unpooled t-test (variance ratio of 8.2)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.011, t-test, 1 sided; Unpooled t-test (variance ratio of 4.7)

36. Post Hoc Outcome: Responder Analysis (≥100%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline and with the ability to maintain fixation at Baseline (N=42), with a responder being defined as someone who gains at least 100% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: Per Protocol (PP) Population with ≤15 letter baseline BCVA disparity between eyes and ability to maintain fixation - 41 subjects from this population completed the study, of which 37 posted a measurable CS value at both baseline and 12 months. Missing values were not imputed for purposes of this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 13 | 11 | 13
Participants | 0 | 2 | 5
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.039, Fisher Exact

37. Post Hoc Outcome: Responder Analysis (≥150%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline and with the ability to maintain fixation at Baseline (N=42), with a responder being defined as someone who gains at least 150% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 13 | 11 | 13
Participants | 0 | 0 | 4
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.096, Fisher Exact

38. Post Hoc Outcome: Responder Analysis (≥200%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye at baseline and with the ability to maintain fixation at Baseline (N=42), with a responder being defined as someone who gains at least 200% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 13 | 11 | 13
Participants | 0 | 0 | 2
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.480, Fisher Exact

39. Post Hoc Outcome: Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. The data shown here are for mean change from baseline to 12 months in the peak of the CS curve in the PP Population with a study eye that is ≤15 letters worse than the fellow eye and with the ability to maintain fixation at Baseline (N=42). Refer to Outcome Measure #16 for background information on this analysis population. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Peak CS
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 13 | 11 | 13
Peak CS | 0.812 (2.049) | 0.020 (2.877) | 7.089 (14.703)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.076, t-test, 1 sided; Unpooled t-test (variance ratio of 51.5)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.057, t-test, 1 sided; Unpooled t-test (variance ratio of 26.1)

40. Post Hoc Outcome: Kinetic Visual Field (KVF) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: Mean change in total area (degrees squared) of all islands of vision from baseline to 12 months in the Per Protocol (PP) Population with a study eye that is ≤15 letters worse than the fellow eye and with the ability to maintain fixation at baseline (N=42). Refer to Outcome Measure #16 for background information on this analysis population.
Time Frame: 12 months
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Total area (degrees squared)
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 14 | 14 | 13
Total area (degrees squared) | 135.14 (595.55) | -94.83 (1039.37) | 1263.68 (3208.76)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.117, t-test, 1 sided; Unpooled t-test (variance ratio of 29.0)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.083, t-test, 1 sided; Unpooled t-test (variance ratio of 9.5)

41. Post Hoc Outcome: Low Luminance Mobility Test (LLMT) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: The LLMT identifies the performance of RP patients as they walk along an indoor pathway of arrows and obstacles at varying lighting levels. The Critical Illumination Level (CIL) is the light level below which the patient has a markedly slower pace and more errors than all light levels above (brighter than) that point. The LLMT uses light levels that go from very dim (0.12 lux) to very bright (500 lux), with evenly spaced increments that increase light by doubling the brightness of the room from the prior level. These evenly spaced light levels have been converted to a scale score to enable easier calculation of change scores. The dimmest level of 0 lux corresponds to a scale score of 13, whereas the brightest level of 500 lux corresponds to a scale score of 0. A positive scale score change from baseline to 12 months represents improvement, whereas a negative scale score change represents a decline. Refer to Outcome Measure #16 for background information on this analysis population.
Time Frame: 12 months
Population: Per Protocol (PP) Population with ≤15 letter baseline BCVA disparity between eyes and ability to maintain fixation - 41 subjects from this population completed the study, of which 38 posted a measurable CIL value at both baseline and 12 months. Missing values were not imputed for purposes of this analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 12 | 13 | 13
scores on a scale | 0.33 (0.78) | 0.23 (1.01) | 0.92 (2.02)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.172, t-test, 1 sided; Unpooled t-test (variance ratio of 6.7)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.140, t-test, 1 sided; Pooled t-test (variance ratio of 3.98)

42. Post Hoc Outcome: Low Vision Functional Questionnaire (Mobility) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes & Ability to Maintain Fixation
Description: as for outcome 19
Time Frame: 12 months
Population: Per Protocol (PP) Population with ≤15 letter baseline BCVA disparity between eyes and ability to maintain fixation - 41 subjects from this population completed the study. Missing values were not imputed for purposes of this analysis.
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 14 | 14 | 13
logits | -0.054 (0.412) | 0.237 (0.306) | 0.676 (0.957)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.011, t-test, 1 sided; Unpooled t-test (variance ratio of 5.4)

43. Post Hoc Outcome: Responder Analysis (≥10 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21), with a responder being defined as someone who gains at least 10 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. Central foveal thickness, as measured by optical coherence tomography (OCT), is believed to be an anatomical marker representing the number of surviving foveal cones. A thicker central fovea corresponds to more surviving cone photoreceptors which are available to be up-regulated.
Time Frame: 12 months
Population: Per Protocol (PP) Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 8 | 5 | 8
Participants | 1 | 1 | 6
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.0406, Fisher Exact

44. Post Hoc Outcome: Responder Analysis (≥13 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21), with a responder being defined as someone who gains at least 13 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. Central foveal thickness, as measured by optical coherence tomography (OCT), is believed to be an anatomical marker representing the number of surviving foveal cones. A thicker central fovea corresponds to more surviving cone photoreceptors which are available to be up-regulated.
Time Frame: 12 months
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 8 | 5 | 8
Participants | 0 | 1 | 6
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.007, Fisher Exact

45. Post Hoc Outcome: Responder Analysis (≥15 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21), with a responder being defined as someone who gains at least 15 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. Central foveal thickness, as measured by optical coherence tomography (OCT), is believed to be an anatomical marker representing the number of surviving foveal cones. A thicker central fovea corresponds to more surviving cone photoreceptors which are available to be up-regulated.
Time Frame: 12 months
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 8 | 5 | 8
Participants | 0 | 1 | 5
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.026, Fisher Exact

46. Post Hoc Outcome: Responder Analysis (≥20 Letters): Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21), with a responder being defined as someone who gains at least 20 letters in BCVA (assessed by E-ETDRS) from baseline to month 12. Central foveal thickness, as measured by optical coherence tomography (OCT), is believed to be an anatomical marker representing the number of surviving foveal cones. A thicker central fovea corresponds to more surviving cone photoreceptors which are available to be up-regulated.
Time Frame: 12 months
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 8 | 5 | 8
Participants | 0 | 0 | 3
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.200, Fisher Exact

47. Post Hoc Outcome: Best Corrected Visual Acuity (BCVA) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Mean change in BCVA in study eye from baseline to month 12 as assessed by E-ETDRS in the Per Protocol (PP) population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21). Central foveal thickness, as measured by optical coherence tomography (OCT), is believed to be an anatomical marker representing the number of surviving foveal cones. A thicker central fovea corresponds to more surviving cone photoreceptors which are available to be up-regulated. Refer to Outcome Measure #1 for more information on how change in BCVA from baseline to month 12 is assessed.
Time Frame: 12 months
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Letters correct
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 8 | 5 | 8
Letters correct | 3.50 (3.96) | -0.40 (10.36) | 18.38 (18.68)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.030, t-test, 1 sided; Unpooled t-test (variance ratio of 22.2)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.033, t-test, 1 sided; Pooled t-test (variance ratio of 3.3)

48. Post Hoc Outcome: Responder Analysis (≥100%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) Population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21), with a responder being defined as someone who gains at least 100% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: Per Protocol (PP) Population ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness - all 21 subjects from this population completed the study, of which 19 posted a measurable CS value at both baseline and 12 months. Missing values were not imputed for purposes of this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 7 | 4 | 8
Participants | 0 | 0 | 3
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.200, Fisher Exact

49. Post Hoc Outcome: Responder Analysis (≥150%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) Population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21), with a responder being defined as someone who gains at least 150% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 48
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 7 | 4 | 8
Participants | 0 | 0 | 3
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.200, Fisher Exact

50. Post Hoc Outcome: Responder Analysis (≥200%): Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Comparison of responder rates across treatment groups in the Per Protocol (PP) Population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21), with a responder being defined as someone who gains at least 200% in Peak CS from baseline to month 12. Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 48
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 7 | 4 | 8
Participants | 0 | 0 | 1
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 1, Fisher Exact

51. Post Hoc Outcome: Peak Contrast Sensitivity (CS) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Assessment of the ability to detect changes in shades of grey, as measured with a vertical striped pattern that varies in width (cycles per degree or CPD); CS thresholds are created by taking the mean of multiple trials at each pattern width. A CS curve is created using a minimum of three pattern widths, one at the subject's peak or highest sensitivity, and then one larger and smaller pattern width on either side of the peak. The data shown here are for mean change from baseline to 12 months in the peak of the CS curve in the Per Protocol (PP) Population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at baseline (N=21). Refer to Outcome Measure #24 for background information on this analysis population. Refer to Outcome Measure #2 for more information on how change in CS from baseline to 12 months is assessed.
Time Frame: 12 months
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Peak CS
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 7 | 4 | 8
Peak CS | 0.777 (0.732) | -1.343 (2.492) | 10.791 (18.018)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.080, t-test, 1 sided; Unpooled t-test (variance ratio of 606.4)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.050, t-test, 1 sided; Unpooled t-test (variance ratio of 52.3)

52. Post Hoc Outcome: Kinetic Visual Field (KVF) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: Mean change in total area (degrees squared) of all islands of vision from baseline to 12 months in the Per Protocol (PP) Population with a study eye that is ≤15 letters worse than the fellow eye, the ability to maintain fixation, and with at least 130µm of central foveal thickness (as measured in the central subfield region) remaining at bbaseline (N=21). Refer to Outcome Measure #24 for background information on this analysis population.
Time Frame: 12 months
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Total area (degrees squared)
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 8 | 5 | 8
Total area (degrees squared) | 393.93 (613.69) | 107.50 (873.65) | 2251.86 (3668.83)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.099, t-test, 1 sided; Unpooled t-test (variance ratio of 35.7)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.076, t-test, 1 sided; Unpooled t-test (variance ratio of 17.6)

53. Post Hoc Outcome: Low Luminance Mobility Test (LLMT) - PP Population With ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness
Description: The LLMT identifies the performance of RP patients as they walk along an indoor pathway of arrows and obstacles at varying lighting levels. The Critical Illumination Level (CIL) is the light level below which the patient has a markedly slower pace and more errors than all light levels above (brighter than) that point. The LLMT uses light levels that go from very dim (0.12 lux) to very bright (500 lux), with evenly spaced increments that increase light by doubling the brightness of the room from the prior level. These evenly spaced light levels have been converted to a scale score to enable easier calculation of change scores. The dimmest level of 0 lux corresponds to a scale score of 13, whereas the brightest level of 500 lux corresponds to a scale score of 0. A positive scale score change from baseline to 12 months represents improvement, whereas a negative scale score change represents a decline. Refer to Outcome Measure #24 for background information on this analysis population.
Time Frame: 12 months
Population: Per Protocol (PP) Population with ≤15 Letter Baseline BCVA Disparity Between Eyes, Ability to Maintain Fixation, and >130µm Central Foveal Thickness - all 21 subjects from this population completed the study, of which 20 posted a measurable CIL value at both baseline and 12 months. Missing values were not imputed for purposes of this analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
Number analyzed (Participants) | 7 | 5 | 8
scores on a scale | 0.43 (0.98) | -0.60 (0.55) | 1.50 (2.07)
Statistical Analysis 1: Comparison: Sham Treated Control vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.1099, t-test, 1 sided; Unpooled t-test (variance ratio of 4.5)
Statistical Analysis 2: Comparison: Test (jCell Injection) Dose Level 1 vs Test (jCell Injection) Dose Level 2; Test type: Superiority; p = 0.012, t-test, 1 sided; Unpooled t-test (variance ratio of 14.3)

ADVERSE EVENTS:
Time Frame: one year
Groups:
- Sham Treated Control: Mock injection: pressing the hub of a syringe with no needle against the study eye
Arm/Group | Sham Treated Control | Test (jCell Injection) Dose Level 1 | Test (jCell Injection) Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/27 | 0/27
Other Adverse Events (participants affected / at risk) | 13/29 | 18/27 | 14/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Treated Control (N=29) | Test (jCell Injection) Dose Level 1 (N=27) | Test (jCell Injection) Dose Level 2 (N=27)
ocular hypertension (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Treated Control (N=29) | Test (jCell Injection) Dose Level 1 (N=27) | Test (jCell Injection) Dose Level 2 (N=27)
Anterior chamber flare (Eye disorders) | 0 (0) | 0 (0) | 3 (3)
Chalazion (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctival hemorrhage (Eye disorders) | 5 (5) | 9 (9) | 6 (6)
Cystoid macular edema (Eye disorders) | 1 (1) | 2 (3) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 5 (6) | 1 (1)
Visual acuity reduced (Eye disorders) | 3 (3) | 4 (4) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 4 (4) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT03073733/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03073733/SAP_001.pdf